CLINICAL TRIAL: NCT07006181
Title: Effectiveness of Cyproheptadine Hydrochloride Against Appetite to Improve Children's Nutritional Status
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Aryono Hendarto, Head of Doctoral Program in Nutritional Sciences, Principal Investigator, Clinical Professor, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 24081215
Record Dates: First submitted 2025-05-17; First posted 2025-06-05 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Appetite Loss
Keywords: Cyproheptadine hydrochloride; appetite loss; children; mild malnutrition
MeSH Terms: conditions — Anorexia | interventions — Cyproheptadine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cyproheptadine hydrochloride (Experimental): Giving Cyproheptadine hydrochloride dossage 0.25 mg/kg/day divided by 2 dose every 12 hours for 4 weeks.
  Interventions: Drug: cyproheptadine hydrochloride
- Control group (Placebo Comparator): Giving placebo and divided by 2 dose every 12 hours for 4 weeks.
  Interventions: Other: Giving placebo divided by 2 dose every 12 hours for 4 weeks.

INTERVENTIONS:
Drug: cyproheptadine hydrochloride — Giving Cyproheptadine hydrochloride 0.25 mg/kg/day divided by 2 dose every 12 hours for 4 weeks.
  Arms: Cyproheptadine hydrochloride
Other: Giving placebo divided by 2 dose every 12 hours for 4 weeks. — Giving placebo divided by 2 dose every 12 hours for 4 weeks.
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to learn about the benefits of Cyproheptadine hydrochloride in increasing appetite as well as its effect on weight gain in children aged 1-5 years who have difficulty eating. The main questions it aims to answer are:

* Is Cyproheptadine hydrochloride useful in increasing appetite in children?
* Is the Cyproheptadine hydrochloride dose given effective and efficient regarding the improvement of a child's appetite? Can giving Cyproheptadine hydrochloride improve nutritional status of children?
* How long can Cyproheptadine hydrochloride be given to increase appetite in children and what are the side effects?

Participants will:

* Take the Cyproheptadine hydrochloride every day, twice a day for 4 weeks (intervention group); take the placebo (control group)
* Have their ECAST score (score for measuring appetite in children), anthropometric measurement before and after intervention at the second visit (2 weeks), third visit (4 weeks and stop intervention), and fourth visit (8 weeks after stopping the intervention)

DETAILED DESCRIPTION:
This study was conducted in a hospital in the Jakarta region, RS Citra Arafiq. All patients who met the inclusion criteria and had informed consent will be assessed for appetite scoring (ECAST) by the research team and diet analysis as a patient baseline before conducting research. Scoring of appetite and daily calorie achievement was carried out by the team researcher. All patients underwent anthropometric measurements (body weight, height) carried out by the team.

The intervention was carried out for 4 weeks, divided into two groups randomly. During the intervention, caregivers are asked to carry out daily observations and recordings regarding food intake (food records) and weighing 2nd week, 4th week and 8th week. Every patient who meets the inclusion criteria receives education regarding correct feeding rules. Data taken will be analyzed using IBM Statistical Product and Service Solutions (SPSS).

ELIGIBILITY:
Inclusion criterias:

1. Experiencing decreased appetite and/or difficulty eating
2. Poor nutritional status and/or weight faltering
3. The parents agree to participate in the research by signing an informed consent.
4. Patients have National Health Insurance or other health insurance.

Exclusion criterias:

1. Major congenital abnormalities
2. CNS disorders (Cerebral palsy)
3. Inborn errors of metabolism (IEM)
4. GERD (Gastro esophageal reflux disease)
5. Severe acute malnutrition

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2024-11-04 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
ECAST children's appetite scoring | From enrollment, then 4 weeks to the end of treatment at 8 weeks
  ECAST children's appetite questionnaire parameters have been modified into 16 questions and have been validated and implemented. This instrument is about a child's appetite ask most parents or caregivers understand the child's condition at all times. The results of this questionnaire will compared with the average daily calorie achievement. Responses to this instrument were coded as: 1 for "never", 2 for "sometimes" and 3 for "often". The total ECAST score is obtained by summing the responses and a higher score indicates a greater appetite.

SECONDARY OUTCOMES:
Anthropometric status | From enrollment, then 4 weeks to the end of treatment at 8 weeks
  The patient's nutritional status is based on the patient's body weight ratio in kilograms to height in centimeters at when collecting research data, according to the standard deviation value WHO 2006 growth curve in weight for length type according to gender. Weighing weight and height using digital scales and infantometer/stadiometer.
Calorie intake | From enrollment, then 4 weeks to the end of treatment at 8 weeks
  The average number of calories achieved by the children was compared with the child's calorie needs per day.

CONTACTS AND LOCATIONS:
Locations (1):
- Citra Arafiq Hospital, Jakarta, Indonesia